CLINICAL TRIAL: NCT06272643
Title: Comparison Between Optical Coherence Tomography and Intravascular Ultrasound for Intermediate Left Main Coronary Artery Lesions
Acronym: EMPERATRIZ
Status: Active, not recruiting | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: EPIC36-EMPERATRIZ
Record Dates: First submitted 2024-02-01; First posted 2024-02-22 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Coronary Disease
Keywords: Left main coronary artery; Percutaneous coronary intervention; Intravascular ultrasound; Optical coherence tomography
MeSH Terms: conditions — Coronary Disease | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Left Main Coronary Artery lesion (25-60%)
  Interventions: Diagnostic Test: IVUS (Intravascular Ultrasound) and OCT (Optical Coherence Tomography)

INTERVENTIONS:
Diagnostic Test: IVUS (Intravascular Ultrasound) and OCT (Optical Coherence Tomography) — OCT and IVUS in Patients with LMCA lesion (25-60%)

SUMMARY:
Significant coronary disease of the left main coronary artery (LMCA) is found in 4%-5% of all coronary angiography procedures. Classically, it has been determined that a significant angiographic stenosis should reach at least 50% of the vessel diameter by visual estimation, which corresponds to 75% of the vessel area. However, angiography has a number of limitations inherent to the technique and location of stenosis, and other techniques are therefore available for evaluation. Intracoronary ultrasound (IVUS) deserves, together with the pressure guidewire, special consideration in determining the severity assessment (anatomical and functional) of lesions in this location. Using IVUS the most commonly used cut-off value is 6 mm2. in ambiguous lesions of the LMCA, a MLA >6 mm2 would indicate no revascularisation, a MLA <4.5-5 mm2 would indicate revascularisation, and MLA values between 4.5-5 and 6 mm2 would make it advisable to use FRF/iFR to decide. Optical coherence tomography (OCT) is another intracoronary imaging modality, with greater resolution and significant differences from IVUS. no MLA cut-off point with OCT has been demonstrated for the management of LMCA lesions. Due to the differences in imaging with both techniques, the thresholds established as cut-off points in IVUS cannot be extrapolated to OCT. The objective is to compare the minimal luminal area by IVUS and OCT of angiographically intermediate LCMA lesions and to assess the prognostic value of TCFA assessed by OCT.

DETAILED DESCRIPTION:
Significant coronary disease of the left main coronary artery (LMCA) is found in 4%-5% of all coronary angiography procedures. It is a particularly important site, since it supplies up to 75% of myocardial blood supply, and damage at this level thus implies a large amount of left ventricular myocardium at risk, with a mortality rate close to 40% at 3 years, if revascularisation is not performed.

Anatomically, it has a number of particularities compared to the rest of the coronary arteries, such as its larger diameter (5±0.5 mm) and variable length (10.5±5.3 mm), a composition, particularly at the aorto-ostial level, more similar to the aorta than to the coronary arteries, and in up to 20-30% of the population there is also a division between the anterior descending artery (LAD) and the circumflex artery (LCx) of a third branch called the ramus intermedius or bisector branch.

Classically, it has been determined that a significant angiographic stenosis should reach at least 50% of the vessel diameter by visual estimation, which corresponds to 75% of the vessel area. However, angiography has a number of limitations inherent to the technique and location of stenosis, and other techniques are therefore available for evaluation. Intracoronary ultrasound (ICUS or IVUS) deserves, together with the pressure guidewire, special consideration in determining the severity assessment (anatomical and functional) of lesions in this location.

Several ICUV studies have attempted to find a minimum luminal area (MLA) as the cut-off point, ranging from 4.5-7.5 mm2, to decide whether to perform revascularisation or not. However, the most commonly used cut-off value is 6 mm2 for various reasons. First, it is correlated with functionally significant values using pressure guidewire. Second, the linear law is applied (assuming the fractal nature of the vasculature and a cut-off value of 3 mm2 for the LMCA branches). Finally, it has been validated by the prospective LITRE study with clinical results at 2 years of follow-up. Other studies in Asian population have proposed lower cut-off values (4.5 mm2). However, this population has different body size and therefore smaller LMCA size, the study has lower sensitivity (1/4 of patients with area >4.5 mm2 had positive pressure guidewire), and clinical validation is not presented unlike the LITRE study.

In addition to its value in diagnosis, use of ICUSE allows for optimisation of percutaneous coronary intervention (PCI) if necessary, with decreased events as compared to angiography. Therefore, current clinical practice guidelines consider the use of IVUS to stratify the severity of all LMCA lesions as an indication IIa B. In turn, it has been proposed to integrate the use of ICUS and pressure guidewire in the assessment of doubtful LMCA lesions. Thus, in ambiguous lesions of the LMCA, a MLA >6 mm2 would indicate no revascularisation, a MLA <4.5-5 mm2 would indicate revascularisation, and MLA values between 4.5-5 and 6 mm2 would make it advisable to use FRF/iFR to decide.

Optical coherence tomography (OCT) is another intracoronary imaging modality, with greater resolution and significant differences from ICUS. It is an expanding technique. However, its usefulness in LMCA is somewhat more limited, mainly due to the difficult technique of complete filling with contrast and the native area of the ostial segments. Another disadvantage of its use in LMCA is its limited penetration depth (2-3 mm) compared to ICUS (4-8 mm), and since the LMCA usually has diameters of 3.5-4.5 mm, inadequate assessment may occur. In addition, no MLA cut-off point with OCT has been demonstrated for the management of LMCA lesions. On the other hand, because of the differences in imaging with both techniques, the thresholds established as cut-off points in IVUS cannot be extrapolated to OCT. There are, however, some correlation studies between ICUS and OCT, both in vivo and in vitro, but not specifically in LMCA. In all these studies, it has been shown that ICUS consistently overestimates OCT measurement by ≈10%, the latter being the closest to the real value. The underuse of this technique in the LCMA is justified by the potential technical problems already mentioned and the lack of a validated MLA cut-off point at this level. The potential prognostic implication of finding, even in patients with functionally nonsignificant lesions, vulnerable plaques or thin-cap fibroatheromas (TCFAs) in OCT has recently been highlighted. The objective is to compare the minimal luminal area by ICUS and OCT of angiographically intermediate LCMA lesions and to assess the prognostic value of TCFA assessed by OCT.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years
* Patients with intermediate lesion in the LMCA (Left Main Coronary Artery) (25-60% angiographic stenosis by visual estimation) in whom a study with intracoronary imaging technique is considered (at least one pullback with IVUS (Intravascular ultrasound) and OCT (OPTICAL COHERENCE TOMOGRAPHY) from one of the main branches is mandatory).
* Patients able to give informed consent form.

Exclusion Criteria:

* Patients with indication for coronary surgery regardless of significance of LMCA lesion.
* Patients with LMCA lesion showing ulceration, dissection or thrombus.
* Patients with lesion in a previous functioning arterial or venous graft in the territory supplied by the LMCA (protected LMCA).
* Patients with acute coronary syndrome with potentially culpable injury in LMCA.
* Patients unable to give informed consent.
* Patients with ostial LMCA lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intermediate lesion in the LMCA (Left Main Coronary Artery) (25-60% angiographic stenosis by visual estimation) in whom a study with intracoronary imaging technique is considered (at least one pullback with IVUS (Intravascular ultrasound) and OCT (OPTICAL COHERENCE TOMOGRAPHY) from one of the main branches is mandatory)
Sampling Method: Non-Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
To assess the agreement between minimum luminal area measured by IVUS and OCT in intermediate LCMA lesions | During intervention
  To assess the agreement between minimum luminal area measured by IVUS and OCT in intermediate LCMA lesions in patients with PCI for MLA in ICUS <6 mm2 and OCT without TCFA.

SECONDARY OUTCOMES:
Cardiac Death | 12 months
  Cardiac Death
Cardiovascular Death | 12 months
  Cardiovascular Death
Acute myocardial infarction of treated/functionally assessed lesion | 12 months
  Acute myocardial infarction of treated/functionally assessed lesion
Acute myocardial infarction of any lesion | 12 months
  Acute myocardial infarction of any lesion
Need for revascularisation of lesion treated/functionally assessed | 12 months
  Need for revascularisation of lesion treated/functionally assessed
Need for revascularisation of any lesion | 12 months
  Need for revascularisation of any lesion
Secondary efficacy endpoint: Clear Image Length | During intervention
  The cumulative length of the OCT pullback containing clear cross-sectional image frames according to the measures used for OCT approval. Corelab Ultreon.
Extend of detectable EEL in LM | During intervention
  To measure the extend of detectable external elastic lamina (EEL) in left main artery (LM) with the corelab ultreon software, defined by length in mm and circunferencial grades (up to 360º) of EEL
Correlation between contrast volume used and results, as well as the average contrast volume used in the study. | 30 days after intervention
  Correlation between contrast flow and total volume used and results, as well as the average contrast volume used in the study. The contrast flow and total volume would be expresed in ml/sec and ml respectively, and results will be determinated in the corelab with the ultreon software as interpretable images or not interpretable images. The average contrast volume in ml, will be correlated with the incidence of contrast induced nephropathy defined as the impairment of kidney function-measured as either a 25% increase in serum creatinine (SCr) from baseline or a 0.5 mg/dL (44 µmol/L) increase in absolute SCr value-within 48-72 hours after intravenous contrast administration.

CONTACTS AND LOCATIONS:
Locations (18):
- Spain (18):
  - Hospital General Universitari Dr Balmis, Alicante
  - Hospital Clinico San Carlos, Aravaca
  - Hospital Universitari Vall Hebron, Barcelona
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario de Cabueñes, Gijón
  - Hospital Universitario Juan Ramon Jimenez, Huelva
  - Hospital Universitario de Jerez de La Frontera, Jerez de la Frontera
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de Leon, León
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clinico Universitario de Valladolid, Valladolid
  - Hospital Universitario Lozano Blesa, Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M. 'Ten commandments' for the 2018 ESC/EACTS Guidelines on Myocardial Revascularization. Eur Heart J. 2019 Jan 7;40(2):79-80. doi: 10.1093/eurheartj/ehy855. No abstract available. PMID 30615155
- [Background] de la Torre Hernandez JM, Hernandez Hernandez F, Alfonso F, Rumoroso JR, Lopez-Palop R, Sadaba M, Carrillo P, Rondan J, Lozano I, Ruiz Nodar JM, Baz JA, Fernandez Nofrerias E, Pajin F, Garcia Camarero T, Gutierrez H; LITRO Study Group (Spanish Working Group on Interventional Cardiology). Prospective application of pre-defined intravascular ultrasound criteria for assessment of intermediate left main coronary artery lesions results from the multicenter LITRO study. J Am Coll Cardiol. 2011 Jul 19;58(4):351-8. doi: 10.1016/j.jacc.2011.02.064. PMID 21757111
- [Background] Wang Y, Mintz GS, Gu Z, Qi Y, Wang Y, Liu M, Wu X. Meta-analysis and systematic review of intravascular ultrasound versus angiography-guided drug eluting stent implantation in left main coronary disease in 4592 patients. BMC Cardiovasc Disord. 2018 Jun 14;18(1):115. doi: 10.1186/s12872-018-0843-z. PMID 29898668
- [Background] Kubo T, Akasaka T, Shite J, Suzuki T, Uemura S, Yu B, Kozuma K, Kitabata H, Shinke T, Habara M, Saito Y, Hou J, Suzuki N, Zhang S. OCT compared with IVUS in a coronary lesion assessment: the OPUS-CLASS study. JACC Cardiovasc Imaging. 2013 Oct;6(10):1095-1104. doi: 10.1016/j.jcmg.2013.04.014. Epub 2013 Sep 4. PMID 24011777
- [Background] Kedhi E, Berta B, Roleder T, Hermanides RS, Fabris E, IJsselmuiden AJJ, Kauer F, Alfonso F, von Birgelen C, Escaned J, Camaro C, Kennedy MW, Pereira B, Magro M, Nef H, Reith S, Al Nooryani A, Rivero F, Malinowski K, De Luca G, Garcia Garcia H, Granada JF, Wojakowski W. Thin-cap fibroatheroma predicts clinical events in diabetic patients with normal fractional flow reserve: the COMBINE OCT-FFR trial. Eur Heart J. 2021 Dec 1;42(45):4671-4679. doi: 10.1093/eurheartj/ehab433. PMID 34345911